## **Evaluation of Data**

Statistical Package for the Social Sciences 22.0 (SPSS) computer program will be used to evaluate the data.

The data will be evaluated in the SPSS 22.0 package program.

- In order to determine which method will be used in the analysis of the data, the normal distribution of the groups will be decided by checking the Shapiro-Wilk, Kolmogorov-Smirnov conformity, kurtosis and skewness values. Analysis results will be displayed as percentage, mean and standard deviation.
- T-test for difference between two independent groups, Anova test will be used to compare difference between more than two groups. Post-Hoc Scheffe and Tukey tests will be used to determine from which group the difference in the results obtained from the Anova test originates.
- The homogeneity of the variance will be determined by looking at the Levene statistics.
- Pearson correlation analysis and linear regression analysis will be performed in order to evaluate the relationship between variables.
- The significance level of p<0.05 will be used as a criterion in the findings.